CLINICAL TRIAL: NCT07329491
Title: Evaluation of the Impact of a Structural Educational Intervention on the Prevention of Diabetic Foot Syndrome: A Ramdomized Clinical Trial Using a Mixed Methods Approach
Brief Title: Impact of an Educational Intervention on Ulcer Incidence, Knowledge, Self-Care, and Quality of Life in Diabetic Foot Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, María del Sol Tejeda Ramírez, Investigador Principal, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 24/742-EC_X
Record Dates: First submitted 2025-12-05; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Complications; Diabetes Education; Diabetes Foot Care
Keywords: Diabetic foot; diabetic foot ulcer; health education; self care; quality of life
MeSH Terms: conditions — Diabetes Complications; Diabetic Foot; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured diabetic foot education program (Experimental): Participants attended two structured, group-based educational sessions on diabetic foot prevention based on IWGDF guidelines, delivered by a specialist, including foot self-care, footwear, and risk identification.
  Interventions: Behavioral: Structured education intervention
- Standard podiatry care without structured education (Active Comparator): Participants received standard care during routine chiropody consultations at a specialised unit, without additional structured educational intervention.
  Interventions: Other: Standard podiatry care

INTERVENTIONS:
Behavioral: Structured education intervention — Participants in the intervention arm received a structured educational program delivered face-to-face in small groups by a healthcare professional specialized in diabetic foot prevention. The program comprised two monthly sessions (2 hours each) following IWGDF recommendations. Session topics included diabetic foot pathophysiology, ulcer risk identification, glycaemic control, daily foot inspection, proper footwear and sock selection, nail care, skin care (hydration/creams) and recognition of warning signs. Teaching methods combined short lectures, visual materials, case examples and group discussion; participants received printed take-home guidance. Knowledge, self-care behaviours and foot skin condition were assessed pre/post intervention and participants were followed for 6 months to monitor outcomes. Structured diabetic foot education.
  Arms: Structured diabetic foot education program
Other: Standard podiatry care — Routine podiatry care provided during regular chiropody consultations at a specialised unit, including clinical foot assessment and usual advice, without any structured or formal educational program.
  Arms: Standard podiatry care without structured education

SUMMARY:
This randomized clinical trial assessed the impact of a structured educational intervention in patients with diabetic foot syndrome. Forty-two participants were allocated to an intervention group-receiving two specialist-led educational sessions-or to a control group with standard care.

The intervention produced significant improvements in knowledge and self-care after the first session, with stable retention and cumulative benefits by the end of the program. Clinically relevant improvements were also observed in skin condition and preventive foot-care behaviors such as appropriate footwear, socks, and nail-cutting technique.

Qualitative data showed that diabetes and DFS strongly affect quality of life, while group-based education enhanced peer support, sense of control, and adherence to preventive care. No ulcers occurred during the six-month follow-up.

Structured educational interventions are effective and rapidly beneficial, though larger studies with longer follow-up are needed to confirm their impact on ulcer prevention.

DETAILED DESCRIPTION:
This randomized clinical trial evaluated the impact of a structured educational intervention on ulcer incidence, patient knowledge, self-care practices, and quality of life in individuals with diabetic foot syndrome (DFS). A total of 42 patients were assigned either to an intervention group-which received two monthly educational sessions delivered by a specialist-or to a control group receiving standard care.

The intervention followed IWGDF recommendations and covered topics such as DFS pathophysiology, glycemic control, ulcer risk identification, and evidence-based preventive strategies. Knowledge was assessed at four time points using a validated questionnaire. Self-care practices were assessed through clinical observation, and skin condition through the CERLCP scale. A qualitative analysis using focus groups explored patients' subjective experiences.

No new foot ulcers developed during the six-month follow-up. The intervention group demonstrated significant improvements in knowledge after the first session, with stable retention between sessions and cumulative gains by the end of the program. Marked improvements were also observed in self-care behaviors, particularly appropriate footwear and socks, nail-cutting technique, and reduction of hyperkeratosis. Skin quality improved with clinically meaningful effect sizes.

The qualitative findings showed that diabetes and DFS substantially affect patients' physical, emotional, social, and economic well-being. The educational intervention enhanced peer support, sense of control, and adherence to preventive self-care.

This study demonstrates that a structured educational intervention-even a single session-can produce rapid and meaningful improvements in knowledge and self-care practices. Larger studies with longer follow-up are required to determine its effectiveness in reducing ulcer incidence over time.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) with a confirmed diagnosis of diabetes mellitus (Type

  1 or Type 2).
* Classified at any risk level for diabetic foot ulceration according to the IWGDF Foot Risk Classification.
* Able to walk independently and capable of participating in educational activities and evaluations.
* Able to understand study procedures and voluntarily provide written informed consent.
* Willing to attend educational sessions (intervention group) and complete all scheduled assessments.

Exclusion Criteria:

* Decline to participate or inability to provide written informed consent.
* Presence of cognitive impairment, neurological disorders, or any condition that limits comprehension or adherence to study procedures.
* Severe physical or functional limitations preventing participation in foot assessments or educational sessions.
* Active diabetic foot ulcer or ongoing treatment for an acute foot wound at enrollment.
* Participation in another clinical trial that could interfere with study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility was determined based on biological sex (male or female), regardless of the participant's gender self-identification.
Enrollment: 42 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of new foot ulceration | Baseline and 6-month follow-up
  Proportion of participants developing a new diabetes-related foot ulcer (yes/no), defined as a full-thickness skin break on the foot. Assessed through clinical examination and medical record review during routine follow-up visits.

SECONDARY OUTCOMES:
Knowledge score (6-item questionnaire) | Baseline, immediately after the first educational session, 30 days later before the second session, and immediately after the second educational session.
  Change in the total score of a validated six-item diabetic foot knowledge questionnaire assessing understanding of diabetic foot pathophysiology, ulcer risk factors, appropriate footwear and sock characteristics, and preventive self-care practices.
  Scale details: The questionnaire consists of 6 dichotomous items (correct/incorrect), with a total score range from 0 to 6 points. Higher scores indicate greater knowledge and a better outcome.
Self-care behaviors (footwear, socks, toenail trimming, orthoses, maceration, hyperkeratosis) | Baseline at the first educational session and immediately after the second educational session, 30 days later.
  Change in individual dichotomous self-care indicators (appropriate footwear, appropriate socks, correct toenail trimming, use of orthoses, interdigital maceration, hyperkeratosis), assessed through direct clinical observation using a standardized checklist.
Sking quality. Questionnaire for the Evaluation of Injury Risk and Skin Quality in Diabetic Foot Sindrome (QERSQ). | Baseline, immediately after the first educational intervention, and immediately after the second educational intervention at 30 days.
  Change in total Questionnaire for the Evaluation of Injury Risk and Skin Quality in Diabetic Foot Sindrome, score evaluating skin condition of the dorsal foot, plantar surface and heel. Higher scores indicate worse skin condition. Score range 0-12
Quality of life related to diabetic foot syndrome (qualitative assessment) | One assessment 30 days after study initiation, immediately following completion of the second educational intervention.
  Qualitative evaluation of quality of life through focus groups, exploring physical, emotional/psychological, social, and economic impact of diabetic foot syndrome, as well as perceived benefits of the structured educational intervention.
  This outcome is qualitative in nature and is not based on a numerical scale or score.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Enfermería, Fisioterapia y Podología de la Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided